CLINICAL TRIAL: NCT06169540
Title: Salivary Extracellular Vesicle Associated lncRNAs in Heart Failure (SEAL-HF)
Acronym: SEAL-HF
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Saumya Das, Director, Resynchronization and Advanced Cardiac Therapeutics Program, Massachusetts General Hospital; Associate Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2022P003352
Record Dates: First submitted 2023-11-16; First posted 2023-12-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: CHF; ADHF; Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Saliva and plasma samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ADHF: Patients with ADHF (during admission and discharge).
- CHF: Patients with CHF.
- Control: Patients undergoing electrophysiology procedures.

SUMMARY:
The purpose of this study is to determine the relationship between the levels of Ribonucleic acid (RNA) circulating molecules, including ones in extracellular vesicles from different organs in the blood and in the saliva of patients with Acute Decompensated Heart Failure (ADHF) and Chronic Heart Failure (CHF) to see if a new, non-invasive diagnostic test can be developed for heart failure exacerbation.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the expression of extracellular vesicle RNAs (evRNAs) during admission for and decongestion of ADHF patients and determine their diagnostic and prognostic potential. The main hypothesis is that these evRNAs are dynamically regulated in response to volume status changes. Thus, the aim is to delineate: i) the utility of salivary evRNA expression in discriminating ADHF from compensated chronic heart failure states in ADHF patients, chronic heart failure patients and controls (n=30 each); and ii) assess changes in expression in ADHF patients during decongestion. Plasma and salivary evRNA levels will be correlated to determine accuracy of salivary Extracellular Vesicles (EVs) to reflect changes in plasma.

This is a multi-cohort study that will make use of clinical saliva and plasma samples of 90 subjects across three groups. The first group will consist of 30 patients admitted to the hospital for ADHF (clinical samples will be collected during acute decompensation and after diuresis of ADHF patients). The second group will consist of 30 patients with chronic heart failure who are seen in the outpatient clinic. The control group will also include 30 patients undergoing electrophysiology procedures recruited through the Electrophysiology Lab (EP). For each group, blood plasma and saliva samples will be obtained.

ELIGIBILITY:
Inclusion Criteria CHF:

* At least 18 years of age
* Stable disease defined as CHF of any type, New York Heart Association (NYHA) functional class II/III/IV, N-terminal pro-B-type natriuretic peptide (NT-proBNP) ≥600 pg/ml if Left Ventricular Ejection Fraction (LVEF) ≤30%; ≥1000 pg/mL if LVEF 31-35%; ≥2500 pg/mL if EF >35%

Inclusion Criteria ADHF:

* At least 18 years of age
* Clinical signs and/or symptoms (including exertional or rest dyspnea, orthopnea or Paroxysmal Nocturnal Dyspnea (PND)) and N-terminal pro-BNP level > 1000 pg/mL or BNP > 400 pg/ml, OR Clinical evidence of congestion: X-ray evidence of pulmonary edema or pleural effusions, elevated Jugular Venous Pulse (JVP), lower extremity edema, or rales on pulmonary examination, right heart catheterization evidence of elevated filling pressures (Right Atrium (RA) pressure > 10 mmHg; Pulmonary Capillary Wedge Pressure (PCWP) > 18 mmHg) and clinical response to Intravenous (IV) diuretic therapy (as judged by a physician)

Inclusion Criteria control:

* At least 18 years of age
* Will/have undergone an EP procedure in the EP lab

Exclusion Criteria:

* Active pregnancy or lactation
* Cardiac amyloidosis
* Active malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve patients admitted to the hospital for ADHF, patients with chronic heart failure who are seen in the outpatient clinic, and control patients recruited through the EP lab.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between weight change (kg), fluid balance (cumulative fluid intake and output, mL), clinical response to diuretic therapy (as judged by a physician), and salivary biomarker levels assessed by quantitative Polymerase Chain Reaction (qPCR) | Through study completion, an average of 1 year
Rehospitalization event prediction | Through study completion, an average of 1 year
  Linear regression analysis for biomarker prediction of subsequent hospital admissions.
Association between known biomarkers (NT-proBNP), volume status (right heart catheterization data, echocardiographic data), and salivary biomarker level assessed by qPCR | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michail Spanos, MD, Study Director — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No